CLINICAL TRIAL: NCT05428345
Title: Post-Marketing Surveillance (Usage Results Study) of Vedolizumab Subcutaneous Injection in Patients With Ulcerative Colitis or Crohn's Disease in South Korea
Brief Title: A Study of Vedolizumab SC Given to Adults With Moderate to Severe Ulcerative Colitis or Crohn's Disease in South Korea
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: VedolizumabSC-4003
Record Dates: First submitted 2022-06-16; First posted 2022-06-23 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Ulcerative Colitis; Crohn's Disease; Inflammatory Bowel Disease (IBD)
Keywords: Drug Therapy
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With UC or CD: Participants diagnosed with moderately to severely active UC and CD, who have had an inadequate response with, lost response to, or were intolerant to either conventional therapy or a TNF-α antagonist and have initiated treatment with vedolizumab in a routine clinical practical setting in South Korea, will be observed prospectively for 52 weeks.

SUMMARY:
The main aim of the study is to observe adult participants in South Korea that are being treated with vedolizumab injected just under the skin (subcutaneous or SC) to treat ulcerative colitis (UC) or Crohn's disease (CD) who have had an in-adequate response with, lost response to, or had too many side effects in response to either conventional therapy or a Tumor Necrosis Factor-alpha (TNF-α) antagonist. This study will observe the side effects and potential benefit to UC and CD participants related to vedolizumab SC treatment with data collection from medical files. There is no treatment involved in this study, this is only an observational review of current collected data relating to adults in South Korea with UC or CD treated with vedolizumab SC.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, post-marketing study of adult participants with moderately to severely active UC or CD, who have had an inadequate response with, lost response to, or were intolerant to conventional therapy or a TNF-α antagonist. This study will evaluate the safety and effectiveness of vedolizumab SC in a routine clinical practice setting under real world condition.

This study will enroll approximately 600 participants. The data will be prospectively collected, at the centers and recorded into electronic case report forms (e-CRFs). All participants will be enrolled in a single observational group:

• Participants with UC or CD

This multi-center trial will be conducted in South Korea. The overall time for data collection in the study will be approximately 6 years.

ELIGIBILITY:
Inclusion Criteria:

1. With moderately to severely active UC or CD, who have had an inadequate response with, lost response to, or were intolerant to either conventional therapy or a TNF-α antagonist
2. With evidence of therapeutic benefit after at least 2 vedolizumab intravenous infusions

Exclusion Criteria:

1. With hypersensitivity such as dyspnea, bronchospasm, urticaria, flushing and increased heart rate to the vedolizumab substance or to any of its excipients
2. With active severe infections such as tuberculosis, cytomegalovirus, sepsis, listeriosis and opportunistic infections such as Progressive Multifocal Leukoencephalopathy (PML)
3. For whom vedolizumab SC is contraindicated as per product label

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll participant with moderately to severely active UC and CD, who have had an inadequate response with, lost response to, or were intolerant to either conventional therapy or a TNF-α antagonist.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Serious Adverse Events (SAEs) | Up to Week 52
Percentage of Participants With Adverse Drug Reactions (ADRs) | Up to Week 52
Percentage of Participants With Serious Adverse Drug Reactions (SADRs) | Up to Week 52
Percentage of Participants With Adverse Events of Special Interest (AESIs) | Up to Week 52
Percentage of Participants With Unexpected Adverse Events (AEs) | Up to Week 52
Percentage of Participants With Unexpected ADRs | Up to Week 52

SECONDARY OUTCOMES:
Percentage of Participants With UC and CD Who Achieved Clinical Response | Up to Week 52
  Clinical response:reduction of Mayo score of greater than or equal to(>=)3points and >=30 percent(%) from baseline score, with an accompanying decrease in rectal bleeding subscore >=1 point/an absolute rectal bleeding sub-score of less than or equal to(<=)1 point in UC participants;and reduction of Crohn's Disease Activity Index (CDAI) score >=70 points from baseline score in CD participants. Total Mayo score measures disease activity of UC;comprise of 4 sections: stool frequency,rectal bleeding,physician rating of disease activity,endoscopic findings. Each graded from 0-3. Total scores range from 0-12.Higher scores indicate more severity.CDAI assesses CD based on clinical signs such as number of liquid stools,abdominal pain,general wellbeing,presence of complications,opiates for diarrhea,presence of abdominal mass, hematocrit. CDAI consist of eight factors,each summed after adjustment with a weighting factor. Total score ranged from 0-600 points.Higher scores indicate more severity.
Percentage of Participants With UC and CD Who Achieved Clinical Remission | Up to Week 52
  Clinical remission is defined as: total Mayo score <=2 and no individual sub-score greater than (>) 1 point in UC participants; and CDAI score less than (<) 150 points in CD participants. Total Mayo score measures disease activity of UC; comprise of 4 sections: stool frequency, rectal bleeding, physician rating of disease activity, endoscopic findings. Each graded from 0-3. Total scores range from 0-12. Higher scores indicate more severity. CDAI assesses CD based on clinical signs such as number of liquid stools, abdominal pain, general wellbeing, presence of complications, opiates for diarrhea, presence of abdominal mass, hematocrit. CDAI consist of eight factors, each summed after adjustment with a weighting factor. Total score ranged from 0-600 points. Higher scores indicate more severity.
Percentage of Participants With UC and CD Who Achieved Mucosal Healing | Up to Week 52
  Mucosal healing is defined as: Mayo endoscopic sub-score of <=1 point in the UC participants; and Crohn's Disease Endoscopic Index of Severity (CDEIS) score <3.5 points in the CD participants. Mayo score: instrument to measure disease activity of UC; consists of 4 variables: stool frequency, rectal bleeding, physician rating of disease activity, and endoscopic findings. Each graded from 0-3. Total score range of 0-12. Higher scores indicating more severity. CDEIS comprise of 4 sections assessing endoscopic severity of CD in 5 segments: rectum; sigmoid and left colon; transverse colon; right colon; ileum in terms of: deep ulcerations, superficial ulcerations, surface involved by disease and ulcerated surface measured. The presence of ulcerate and non-ulcerated stenosis will be recorded in each segment. CDEIS score range from 0-44 with a higher score indicating greater severity of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- Donggguk University Ilsan Hospital, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language. — https://clinicaltrials.takeda.com/study-detail/52b934f938554c0e?idFilter=%5B%22VedolizumabSC-4003%22%5D